CLINICAL TRIAL: NCT01640704
Title: Impact of Computerized Reminders on Blood Pressure Documentation and Control
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, david bates, Chief, General Internal Medicine, BWH, Agency for Healthcare Research and Quality (AHRQ)
Allocation: Randomized | Model: Factorial | Masking: Double
Other Study IDs: 3Ui8HS11046
Record Dates: First submitted 2012-07-12; First posted 2012-07-16 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

INTERVENTIONS:
Behavioral: Computerized reminders about treatment guidelines to providers who care for hypertensive patients

SUMMARY:
Numerous studies have examined potential causes for the racial differences in HTN prevalence and severity including baseline insulin levels, sympathetic nervous activity, intracellular calcium levels and intracellular sodium levels.[21-23] However, to our knowledge, there have been no studies examining the relationship of physician adherence to JNC guidelines to racial disparities in outcomes from HTN; nor have there been published studies examining the use of interventions such as computerized decision support tools or case-management to improve JNC adherence with the goal of reducing racial differences in blood pressure control. The aims of this study are: 1) To determine if physician's prescribing practices for HTN medications adhere to JNC guidelines for drug therapy.

2) To determine if there are variations in adherence to JNC guidelines based on patient race.

3) To determine if adherence to JNC guidelines improves blood pressure control. 4) To determine if the use of computerized medical reminders improves adherence to JNC guidelines.

ELIGIBILITY:
Inclusion Criteria:

We examined data obtained from the electronic medical record review of patients older than 20 years with a diagnosis of hypertension, with at least one hypertension-related outpatient visit to one of fourteen general medicine clinics in community health centers, community-based practices, and hospital-based practices affiliated with a large urban academic medical center during the one-year period prior to the beginning of the intervention trial.

Exclusion Criteria:

Patients without documented hypertension-related primary care visits or less than 20 years of age

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2003-07; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: LeRoi S. Hicks, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Gandhi TK, Seger AC, Overhage JM, Murray MD, Hope C, Fiskio J, Teal E, Bates DW. Outpatient adverse drug events identified by screening electronic health records. J Patient Saf. 2010 Jun;6(2):91-6. doi: 10.1097/PTS.0b013e3181dcae06. PMID 22130350